CLINICAL TRIAL: NCT01035983
Title: An Open Label Study to Assess the Safety, Tolerability and Efficacy of Frovatriptan in the Prevention of Menstrually Associated Migraine (MAM) Headaches.
Brief Title: Safety and Tolerability of Frovatriptan to Prevention of Menstrually Associated Migraine (MAM) Headaches
Acronym: MAM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Collaborators: Vernalis (R&D) Ltd (Industry)
Responsible Party: John C. Campbell, Director, Medical Affairs, Endo Pharmaceuticals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VML 251-3MAM03
Record Dates: First submitted 2009-12-17; First posted 2009-12-21 (Estimated); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Migraine
Keywords: menstrually associated migraine (MAM), Migraines,Menstrual Migraines, menstrually related migraines
MeSH Terms: conditions — Migraine Disorders; Limb-girdle muscular dystrophy, type 2C | interventions — frovatriptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Frovatriptan 2.5 mg (Experimental): Frovatriptan 2.5 mg tablets administered orally 2 x 2.5 mg twice daily (loading dose) on day 1, followed by 2.5 mg twice daily days 2 to 6.
  Interventions: Drug: Frovatriptan 2.5 mg

INTERVENTIONS:
Drug: Frovatriptan 2.5 mg

SUMMARY:
In this open-label, multi-center study, patients were treated with frovatriptan for a maximum of 12 perimenstrual periods (PMPs). For each PMP, dosing commenced 2 days before the anticipated onset of the menstrual migraine (MM) headache and continued for a total of 6 days. Patients were to take a loading dose of frovatriptan 5 mg (two tablets) twice daily on Day 1, followed by frovatriptan 2.5 mg twice daily on Days 2-6. During the study, patients were to visit the study site a total of 6 times. Efficacy and/or safety assessments were performed at each visit.

DETAILED DESCRIPTION:
This Phase IIIb, open label, multi-centre study evaluated the safety and tolerability of frovatriptan taken by patients for up to 12 perimenstrual periods (PMPs) for the prevention of menstrual migraine (MM). The study required approximately 300 patients to treat 6 PMPs and 100 patients to treat 12 PMPs. To achieve these numbers, 550 patients were to be enrolled into the study. Once enrolled, patients were requested to treat at least 6 PMPs in the first 9 months and 12 PMPs overall. Patients were to remain in the study for a maximum of 15 months or until they had completed the treatment of 12 PMPs, whichever occurred sooner.Patients were to take a loading dose of frovatriptan 5 mg (two tablets) twice daily on Day 1, followed by frovatriptan 2.5 mg twice daily on Days 2-6.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 15 years and over (≥18 years in United Kingdom and South Africa), with at least a 12 month documented history of experiencing migraine according to IHS criteria, including confirmation of a 3 month diary based documented history of MAM.
* An average frequency of MAM in at least two out of three menstrual cycles, within the previous 12 months
* Regular, predictable menstrual periods
* MAM headaches occurring between Day -2 and day +4 of menses
* Able and willing to sign informed consent and to comply with study procedures, including completion of the diary cards.

Exclusion Criteria:

* More than three migraine attacks per month that were not MAM attacks
* A history of myocardial infarction, ischemic heart disease (or presenting with symptoms or signs compatible with ischemic heart disease), coronary vasospasm or peripheral vascular disease
* Significant cerebrovascular disease including basilar or hemiplegic migraine
* Uncontrolled hypertension (SBP >180 mmHg, DBP >95 mmHg)
* Severe hepatic or renal insufficiency
* More than 15 headache days per month, exclusive of migraine headache
* Any other condition or serious illness which, in the opinion of the investigator, would interfere with optimal participation in the study
* A history of clinically relevant allergy, including that to frovatriptan or other triptans
* Pregnant or breast-feeding, or intending to become pregnant or breast-feed during the study period (patients were to be using adequate contraception and have a negative pregnancy test at screening)
* Treatment with another investigational drug within 30 days or 5 half-lives (whichever was longer) before the screening visit
* Any change in their oral contraceptive medication (if applicable) in the 2 months prior to screening, or anticipation of any change during study participation
* Any change in the type or dose of any prophylactic migraine medication in the 2 months prior to screening, or anticipation of any change during study participation
* A history of migraine with aura, according to IHS criteria, and currently treated with a combined oral contraceptive (South Africa only).

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2003-12; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Incidence of all treatment-emergent adverse events (AEs). | 9-15 months

SECONDARY OUTCOMES:
Incidence of menstrual migraine headache | 9-15 months
Maximum headache severity | 9-15 months
Number of headache-free days during a treated perimenstrual period (PMP) | 9-15 months
Occurrence and severity of menstrual migraine headache-associated symptoms | 9-15 months
Maximum functional impairment during menstrual migraine headache | 9-15 months
Incidence and severity of intercurrent migraine | 9-15 months
Total migraine burden | 9-15 months
Standard hematology and biochemistry | 9-15 months
12-lead electrocardiogram (ECG) and vital signs, physical examination | 9-15 months
Short-form 12 (SF-12) Health Related Quality of Life Questionnaire | 9-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Anne MacGregor, DIPM MFFP, Principal Investigator — City of London Migraine Clinic
Locations (5):
- Munich, Germany
- Budapest, Hungary
- Warsaw, Poland
- Cape Town, South Africa
- London, United Kingdom

REFERENCES:
- [Result] MacGregor EA, Brandes JL, Silberstein S, Jeka S, Czapinski P, Shaw B, Pawsey S. Safety and tolerability of short-term preventive frovatriptan: a combined analysis. Headache. 2009 Oct;49(9):1298-314. doi: 10.1111/j.1526-4610.2009.01513.x. PMID 19788471